CLINICAL TRIAL: NCT00651612
Title: Study to Evaluate Safety of Brimonidine/Timolol Fixed Combination in Glaucoma or Ocular Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190342-024T
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Brimonidine Tartrate; Timolol; Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Brimonidine 0.2%/Timolol 0.5% Fixed Combination Ophthalmic Solution
  Interventions: Drug: Brimonidine 0.2%/Timolol 0.5% Fixed Combination Ophthalmic Solution
- 2 (Active Comparator): Concurrent Brimonidine 0.2% and 0.5% Timolol
  Interventions: Drug: Concurrent brimonidine 0.2% and 0.5% timolol

INTERVENTIONS:
Drug: Brimonidine 0.2%/Timolol 0.5% Fixed Combination Ophthalmic Solution — Brimonidine 0.2%/timolol 0.5% fixed combination ophthalmic solution 1 drop instilled in each eye two times daily (morning and evening)
  Other Names: COMBIGAN™
  Arms: 1
Drug: Concurrent brimonidine 0.2% and 0.5% timolol — Brimonidine 0.2%, 1 drop instilled in each eye three times daily (morning, afternoon, and evening) and timolol 0.5% timolol, 1 drop instilled in each eye twice daily (morning and evening) and vehicle of brimonidine combination ophthalmic solution 1 drop instilled in each eye (morning, afternoon and/or evening)
  Arms: 2

SUMMARY:
This study evaluates the safety of brimonidine/timolol fixed combination in glaucoma or ocular hypertension patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ocular hypertension or glaucoma
* Patient requires IOP-lowering therapy in both eyes

Exclusion Criteria:

* Uncontrolled medical conditions
* Contraindication to β-adrenoceptor antagonist therapy or brimonidine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 2005-11; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

REFERENCES:
- See also: Link to Clinical Trial Results — http://www.allerganclinicaltrials.com